CLINICAL TRIAL: NCT03256214
Title: Acute Effects of Open and Closed Suction Systems on Pulmonary Mechanics and Cardiovascular Function in Mechanically Ventilated Patients
Brief Title: Acute Effects of Open and Closed Suction Systems in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 467
Record Dates: First submitted 2017-07-18; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed suction system (Experimental): Patients in mechanical ventilation were aspirated with closed suction system.
  Interventions: Procedure: Closed suction system
- Open suction system (Active Comparator): Patients in mechanical ventilation were aspirated with open suction system.
  Interventions: Procedure: Open suction system

INTERVENTIONS:
Procedure: Closed suction system — In mechanically ventilated patients, intratracheal secretions were aspirated with closed suction systems to compare the pulmonary and cardiovascular parameters (Peak Pressure, Resistance, and Pressure Plateau, Heart Rate and Mean, Diastolic, and Systolic Pressures) with open suction system.
  Arms: Closed suction system
Procedure: Open suction system — In mechanically ventilated patients, intratracheal secretions were aspirated with open suction systems to compare the pulmonary and cardiovascular parameters (Peak Pressure, Resistance, and Pressure Plateau, Heart Rate and Mean, Diastolic, and Systolic Pressures) with closed suction system.
  Arms: Open suction system

SUMMARY:
Seventy-one patients in intensive care were randomized for initial treatment with open suction systems or closed suction systems in a cross-over design. Pulmonary and cardiovascular physiology was assessed immediately before and after three 10-second aspirations per suction. Were analyzed the effect of each suction system on physiologic parameters while adjusting for their respective values prior to suction.

DETAILED DESCRIPTION:
Study Participants. The sample consisted of 71 subjects, both genders, hospitalized in intensive care units. This study protocol was approved by the Research Ethics Committee of Heliopolis Hospital - Sao Paulo - Brazil.

Patients were randomized in the following way: patients hospitalized in the odd beds of ICU were aspirated initially by open suction system (OSS) and later by the closed suction system (CSS); patients hospitalized in the even beds were aspirated by CSS, initially, and subsequently by the OSS.

Cardiopulmonary measures: Eligible patients were evaluated for the presence or absence of neural stimulation to spontaneous ventilation (drive breathing). If the patients showed spontaneous respiratory movements, they were sedated to the level four of Ramsay scale. After this initial evaluation, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), heart rate (HR), respiratory rate (RR), oxygen saturation (SAT), tidal volume (Vt), peak pressure (Ppeak), plateau pressure (Pplat), positive end expiratory pressure (PEEP), and inspiratory flow (V) were measured. The HR and SAT data were collected by visualization of DX 2010 multiparameter monitor from Dixtal. SBP, DBP and MBP were obtained by a single measurement provided by the same monitor. Data of peak pressure, plateau pressure, positive end expiratory pressure, inspiratory flow and tidal volume were used to calculate compliance (C) and airway resistance (R). Data were collected before and after tracheal aspiration.

Pulmonary Suction: After the initial data were obtained, patients who were under volume-controlled ventilation mode (VCV) were submitted to the first aspiration procedure according to randomization described above. Patients who were under pressure-controlled ventilation mode (PCV) were changed to VCV mode, respecting the individual mean tidal volume, which means that the tidal volume of the patient under PCV would be used to ventilate in VCV. All patients were ventilated with a Savina (Drager) mechanical ventilator. Aspiration procedures and data collection were done by a health care professional unaware of the study regimes or objectives. After the measurement of the initial parameters, patients underwent the procedure of aspiration in an open or closed system according to the randomization described above. All patients were aspirated by a system that had not been used previously. The procedure was timed and required 10 seconds to insert and remove the aspiration catheter, with each aspiration performed three times. The outside diameter of the aspiration catheter had half the inner diameter of the endotracheal tube, and the negative pressure was adjusted between 70 and 100 mmHg. At the end of the aspiration procedure, physiological assessments were repeated. Patients were returned to nursing care and underwent the second procedure after six hours from initial aspiration.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old;
* intubated with a 7.5mm endotracheal tube;
* mechanically ventilated.

Exclusion Criteria:

* upper gastrointestinal bleeding;
* hemodynamic instability;
* airway bleeding;
* previous lung diseases.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
Improvements in Pulmonary parameters when comparing closed and open suction systems. | 1 day
  Assessment of Peak Pressure (cmH20) in both closed and open suction systems.
Improvements in Cardiovascular parameters when comparing Closed and open suction systems. | 1 day
  Assessment of Blood Pressure (mmHg) in both closed and open suction systems.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo D Raimundo, Ph.D., Principal Investigator — Faculdade de Medicina do ABC

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raimundo RD, Sato MA, da Silva TD, de Abreu LC, Valenti VE, Riggs DW, Perrow Carll A. Open and Closed Endotracheal Suction Systems Divergently Affect Pulmonary Function in Mechanically Ventilated Subjects. Respir Care. 2021 May;66(5):785-792. doi: 10.4187/respcare.08511. Epub 2021 Mar 9. PMID 33688090